CLINICAL TRIAL: NCT03568292
Title: Effects of Virtual Reality on Pain and Anxiety in Cancer Patients Undergoing Painful Procedures
Brief Title: Virtual Reality in Reducing Pain and Anxiety in Cancer Participants Undergoing Painful Procedures
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting new cohort to open
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virtually Strong, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-17-10; NCI-2018-00759 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-17-10 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I: Virtual Reality (Experimental): Participants receive the VR intervention during bone marrow biopsy or lumbar puncture lasting until completion of the procedure. Participants will be trained to use VR equipment prior to the bone marrow biopsy or lumbar puncture. The headset will cover both eyes with a strap along the back to hold the headset in place. The headset will be attached by a wire to a laptop which will power the headset and provide content. A remote control will be available for assistance in setting up or stopping the content in the case of an event. The VR content will consist of meditation and relaxing techniques through visual and auditory input which can last up to one hour. There will be minimal stimulatory effort to decrease excess movement for the procedure.
  Interventions: Other: Laboratory Biomarker Analysis; Device: Oculus Rift Headset; Other: Questionnaire Administration
- Arm II: No Virtual Reality (Active Comparator): Participants receive standard of care during bone marrow biopsy or lumbar puncture.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II: No Virtual Reality
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Oculus Rift Headset — Subject wears headset for virtual reality intervention during bone marrow biopsy or lumbar puncture procedure
  Arms: Arm I: Virtual Reality
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well virtual reality (VR) works in reducing pain and anxiety in cancer participants undergoing bone marrow biopsy or lumbar puncture. Virtual reality may impact pain and anxiety during and after the procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of VR in patients undergoing procedural intervention.

SECONDARY OBJECTIVES:

I. To estimate differences between the two arms in terms of pain and anxiety. II. To document any adverse events that could possibly be attributed to the VR intervention.

EXPLORATORY OBJECTIVES:

I. Explore the use of biomarkers as a tool to reflect the impact of intervention.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants undergo VR intervention peri-procedure (bone marrow biopsy or lumbar puncture) lasting until completion of the procedure.

ARM II: Participants receive standard of care during procedure (bone marrow biopsy or lumbar puncture).

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with any cancer
* Patient is currently hospitalized and receiving treatment for a primary or secondary cancer at University of Southern California (USC) Norris Comprehensive Cancer Center and Hospital
* Patient is undergoing a bone marrow biopsy or lumbar puncture

Exclusion Criteria:

* Inability to sign informed assent and/or consent
* Patient with an underlying diagnosis of epilepsy, dementia, Parkinson?s disease, primary central nervous system malignancy, brain metastasis, underlying inflammatory or infectious central nervous system disorder, inner ear infection, history of vertigo, baseline visual or hearing impairment, macular degeneration, untreated glaucoma, implantable medical devices or any medical condition that investigator deems contraindicated
* Patient with an underlying chronic pain disorder, anxiety disorder, depressive disorder, or other psychiatric illness unspecified
* Patient with active Clostridium difficile infection
* Patient on any acute (within last < 24 hour [hr]) or chronic pain medication (opioid, nonsteroidal anti-inflammatory drug [NSAID], steroid)
* Patient on chronic steroids > 10 mg prednisone equivalent daily or other immunosuppressant > 1 week
* Patient who is post bone marrow transplant
* Patient with a body mass index (BMI) > 35

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed according to a visual analog scale (VAS) | Up to 1 year
  A visual analogue pain scale is a validated pain measure. A 10 centimeter horizontal line with a 0 (no pain) on the far left and 10 (worst possible pain) on the far right. Participants rate pain intensity by drawing a mark on the line. Pain intensity is obtained by measuring from the 0 to the participant's mark on the line, yielding a score from 0 to 10.
Anxiety | Up to 1 year
  Will be assessed by the State-Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States